CLINICAL TRIAL: NCT02605278
Title: Assessment of a Multicomponent Program for the Integrated Management of Chronic Pain and Depression in Primary Care. Cluster Randomized Clinical Trial
Brief Title: Multicomponent Program for the Integrated Management of Chronic Pain and Depression in Primary Care
Acronym: DROP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI14/00573
Record Dates: First submitted 2015-09-28; First posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-09

CONDITIONS: Depressive Disorder; Musculoskeletal Pain; Chronic Pain
Keywords: Primary Health Care, Patient Education, Care Managament
MeSH Terms: conditions — Depressive Disorder; Musculoskeletal Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical program for pain and depression (Experimental): Structured program with integrated management for depression and chronic musculoskeletal pain with three main components: 1) Optimized care of major depression on the basis of a Clinical Guideline 2) Care Management, and 3) Group psychoeducational intervention.
  Interventions: Other: Clinical program for pain and depression
- Control (Active Comparator): Care as usual
  Interventions: Other: Control

INTERVENTIONS:
Other: Clinical program for pain and depression — Already described
  Other Names: DROP Program (Depression and Pain)
  Arms: Clinical program for pain and depression
Other: Control — Care as usual
  Arms: Control

SUMMARY:
This study evaluates whether the implementation of an integrated clinical program for chronic musculoskeletal pain and depression behave better clinical outcomes than the usual approach in primary care

DETAILED DESCRIPTION:
Chronic musculoskeletal pain and depression are extremely common and relevant pathological conditions, and frequently presented as comorbid processes multiplying the impact on health, worsening the prognosis and complicating the care. The integrated management of both disorders is an opportunity to achieve better clinical outcomes.

AIM: To determinate whether the implementation of an integrated clinical program for chronic musculoskeletal pain and depression behave better clinical outcomes than the usual approach in primary care

METHODS

Design: Cluster randomized clinical trials with two arms:

1. Intervention: Integrated program for depression/chronic pain, and
2. control usual care.

Settings: Primary Care Centers in Tarragona, Spain. Patients: Adults with moderate/severe musculoskeletal pain (Brief Pain Inventory/pain intensity scale > 4 points), with more than three months of evolution and current diagnostic criteria for major depression episode (DSM-IV).

Sample: A total sample of 330 patients (165 control arm and 165 intervention arm) divided into 42 clusters of 8 patients. Cluster composition: patients registered with the same doctor.

Intervention: Structured program with integrated management for depression/ pain with three main components:

1. Optimized care of major depression,
2. Case Management, and
3. Group psychoeducational intervention.

Measurements: "Blind" interviews at 0, 3, 6 and 12 months.

Main outcomes:

* Depressive symptoms (Hopkins Symptom Checklist-20): Severity, response rate and remission rate.
* Pain symptoms (Brief Pain Inventory). Intensity and interference, response rate.
* Disability by psychological problems (Sheehan Disability Inventory)
* Quality of life related to health (EuroQol-5D).

ELIGIBILITY:
Inclusion Criteria:

* Registered patient of a participant doctor
* Chronic musculoskeletal pain moderate to severe (BPI>4), with more than 3 months of duration despite having received analgesic treatment
* Meeting the diagnostic criteria for major depression (DSM IV) at the time of recruitment.

Exclusion Criteria:

* Patients with mental, physical, language limitation or concurrent illness that prevents understanding/participation in the assessments of the study.
* Patients with serious or terminal illness.
* Patients whit psychotic disorder, bipolar disorder or dependence disorder.
* Pregnant or lactating patient
* Patients diagnosed of fibromyalgia or somatization disorder
* Patient in a process of claim for a work disability
* Intervention for a joint prothesis planned forn next 12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Depression severity | 12 months
  Hopkins Symptoms Checklist-Depression HSCL-20
Pain severity | 12 months
  Brief Pain Inventory BPI
Health Related Quality of Life | 12 months
  EuroQol-5D
Pain Interference | 12 months
  Brief Pain Inventory BPI

SECONDARY OUTCOMES:
Depression severity | 3 months
  Hopkins Symptoms Checklist-Depression HSCL-20
Depression severity | 6 months
  Hopkins Symptoms Checklist-Depression HSCL-20
Pain severity | 3 months
  Brief Pain Inventory BPI
Pain severity | 6 months
  Brief Pain Inventory BPI
Health Related Quality of Life | 3 months
  EuroQol-5D
Health Related Quality of Life | 6 months
  EuroQol-5D
Pain Interference | 3 months
  Brief Pain Inventory BPI
Pain Interference | 6 months
  Brief Pain Inventory BPI

CONTACTS AND LOCATIONS:
Overall Officials: Enric Aragonès, MD PhD, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- IDIAP Jordi Gol, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Rambla C, Aragones E, Palleja-Millan M, Tome-Pires C, Lopez-Cortacans G, Sanchez-Rodriguez E, Miro J. Short and long-term predictors of pain severity and interference in primary care patients with chronic musculoskeletal pain and depression. BMC Musculoskelet Disord. 2023 Apr 5;24(1):270. doi: 10.1186/s12891-023-06357-2. PMID 37020278
- [Derived] Aragones E, Rambla C, Lopez-Cortacans G, Tome-Pires C, Sanchez-Rodriguez E, Caballero A, Miro J. Effectiveness of a collaborative care intervention for managing major depression and chronic musculoskeletal pain in primary care: A cluster-randomised controlled trial. J Affect Disord. 2019 Jun 1;252:221-229. doi: 10.1016/j.jad.2019.04.004. Epub 2019 Apr 8. PMID 30986737
- [Derived] Aragones E, Lopez-Cortacans G, Caballero A, Pinol JL, Sanchez-Rodriguez E, Rambla C, Tome-Pires C, Miro J. Evaluation of a multicomponent programme for the management of musculoskeletal pain and depression in primary care: a cluster-randomised clinical trial (the DROP study). BMC Psychiatry. 2016 Mar 16;16:69. doi: 10.1186/s12888-016-0772-2. PMID 27236335